CLINICAL TRIAL: NCT01780181
Title: Randomized Double-blind Controlled Clinical Study of Chemotherapy Combined With or Without Traditional Chinese Medicine on Survival Affect of Elderly Patients With Advanced Non-small-cell Lung Cancer
Brief Title: Clinical Study of Chemotherapy Combined With Chinese Medicine on Survival Affect of Elderly Patients With Lung Cancer
Status: Completed | Type: Observational
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Zhiyi Zhou, Longhua Hospital, Shanghai University of Traditional Chinese Medicine
Other Study IDs: 12401905700zzy
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: lung cancer; traditional Chinese medicine
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — Drug Therapy; Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TCM plus chemotherapy: TCM:oral granules,YangYinFang or YiQiFang or YiQiYangYinFang, four packages,twice a day, three months; Chemotherapy : Intravenous drug use, treated with single-agent chemotherapy :DOC、NVB、GEM.Each cycle was 21-days. Cycles were repeated until disease progression, unacceptable toxicity, or chemotherapy taboo;
  Interventions: Drug: TCM; Drug: Chemotherapy
- Placebo plus chemotherapy: TCM Placebo: oral granules,YangYinFang orYiQiFang or YiQiYangYinFang, 10% of the original dose,four packages,twice a day ,three months; Chemotherapy : Intravenous drug use, treated with single-agent chemotherapy :DOC、NVB、GEM.Each cycle was 21-days. Cycles were repeated until disease progression, unacceptable toxicity, or chemotherapy taboo;
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: TCM — TCM: In China,TCM herbs are given on the basis of the TCM syndrome differentiation as diagnosed by the TCM herbal specialist. Prescriptions formulated into granules origin from Professor Liu Jia-xiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi recipe, benefiting Yin recipe and detoxication and resolving masses recipe.The herbal treatment is adapted to the syndromes.
  Other Names: YangYinFang:four packages twice a day; YiQiFang :four packages twice a day; YiQiYangYinFang:four packages twice a day
  Groups: TCM plus chemotherapy
Drug: Chemotherapy — treated with single-agent chemotherapy :DOC、NVB、GEM DOC 60mg/m2 d1 Q3W NVB 30mg/m2 d1，d8 Q3W GEM 1200mg/m2 d1，d8 Q3W
  Other Names: treated with single-agent chemotherapy :; DOC：Docetaxel; NVB：Vinorelbine; GEM：Gemcitabine

SUMMARY:
The purpose of this study is to observe the efficacy of chemotherapy combined with Traditional Chinese Medicine for elderly patients with advanced non-small-cell lung cancer, also to evaluate the adverse reaction and the reliability.

DETAILED DESCRIPTION:
Non-small-cell lung cancer (NSCLC) accounts for approximately 80% of all lung cancer diagnoses and more than 75% of the patients are diagnosed with an advanced stage. ASCO guidelines recommended that elderly patients with advanced NSCLC use single-agent chemotherapy. Nearly a decade of clinical trials showed that:the median survival time (MST) of Vinorelbine is 5-10months,1-year survival rate is 32%;the MST of Gemcitabine is 6.8-9months,the MST of Taxol is 6.8-10.3months.Research had shown that TCM can prolong long-term survival and improve QOL, but high-level evidence is desperately needed to support this finding.

The investigators perform a multi-center, randomized, double-blind controlled, prospective study in elderly patients with advanced NSCLC. Patients are randomized over observational group (TCM granules plus single-agent chemotherapy), and control group (TCM placebo plus single-agent chemotherapy). The investigators will observe 4 cycles and after that regular follow-up will be arranged. The primary end point is: PFS (progression-free survival); the secondary end points are: (1) OS(overall survival); (2) Objective response rate; (3) TTP(Time-to-Progression); (4) QOL (EORTC QLQ-L43, TCM syndrome score); (5) other end points are: Toxicity, side effects and security of the treatments will be assessed at the same time. The investigators expect that integrated TCM combined with chemotherapy has a better efficacy on prolonging PFS, OS, improving QOL, reducing the adverse reaction of patients than that of chemotherapy.Therefore our study can provide evidences for optimizing and promoting integrated TCM combined with Western Medicine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed of stage IIIb-IV NSCLC ;
2. Ages Eligible for Study: ≥65 years old;
3. Physical status score (ECOG PS) ≤ 2 scores;
4. Estimated life expectancy of at least 12 weeks;
5. Participants have no major organ dysfunction and chemotherapy contraindications: hemoglobin ≥9g/dL, absolute neutrophil count (ANC) ≥1.5*109/L, platelets ≥100 *109/L,bilirubin≤1.5ULN,alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 upper limited number(ULN) (AP, AST, ALT ≤5ULN is acceptable if liver has tumor involvement).INR≤1.5, APTT in the normal range(1.2DLN-1.2ULN),creatinine≤1.5ULN;
6. Informed consent from the patient.

Exclusion Criteria:

1. Patient with other malignant tumor except NSCLC 5 years previous to study entry.
2. Patients who have received single-agent chemotherapy treatment；
3. Estimated life expectancy less than 12 weeks;
4. Serious problem of heart, liver or kidney with severe dysfunction;
5. Pregnant or child breast feeding women;
6. Mental or cognitive disorders;
7. Participating in other drug trials;
8. Who are allergic to the study drug.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Pathologically or cytologically confirmed of stage IIIb-IV NSCLC； Ages Eligible for Study: ≥65 years old; TCM syndromes are deficiency of Yin, deficiency of Qi and deficiency of both Qi and Yin.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | 2 months

SECONDARY OUTCOMES:
overall survival | 2 months
Objective response rate | 2 months
Time-to-Progression(TTP) | 2 months
quality of life(QOL) | one cycle

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyi Zhou, CMD, PhD, Principal Investigator — Longhua Hospital
Locations (1):
- Zhiyi Zhou, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou ZY, Xu L, Li HG, Tian JH, Jiao LJ, You SF, Han ZF, Jiang Y, Guo HR, Liu H. Chemotherapy in conjunction with traditional Chinese medicine for survival of elderly patients with advanced non-small-cell lung cancer: protocol for a randomized double-blind controlled trial. J Integr Med. 2014 May;12(3):175-81. doi: 10.1016/S2095-4964(14)60028-5. PMID 24861837